CLINICAL TRIAL: NCT04396353
Title: The Impact of EXercise TRAining, Physical Activity and Sedentary Lifestyle on Clinical Outcomes in Surviving Patients Infected With the Severe Acute Respiratory Syndrome Coronavirus 2: Cross-sectional Study
Brief Title: EXercise TRAining and Sedentary Lifestyle on Clinical Outcomes in Patients With COVID-19
Acronym: WHO
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; SARS-CoV 2; Corona Virus Infection; Sedentary Behavior
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physically active: Those who receive regular amounts of physical activity. Those who participate in a minimum of 150 minutes of moderate exercise, or 75 minutes of a more vigorous regimen as recommended by the health organizations. Additionally, a person who spend less time sitting (i.e. watching television, surfing the web, playing video games).
  Interventions: Other: Electronic questionnaire
- Sedentary: Those who do not receive regular amounts of physical activity. Where physical inactivity is considered the failure to meet the recommendations of the health organizations, stating that an individual should participate in a minimum of 150 minutes of moderate exercise, or 75 minutes of a more vigorous regimen. Sitting about 70-85% of the time (i.e. watching television, surfing the web, playing video games) is also considered a person living a sedentary lifestyle.
  Interventions: Other: Electronic questionnaire

INTERVENTIONS:
Other: Electronic questionnaire — Clinical, anthropometric, and sociodemographic variables to characterize the sample will be collected using the Google Form. The same tool will be used to collect clinical variables (outcomes), as well as to obtain data on the level of physical activity and sedentary behavior time (predictor variables) prior to SARS-CoV-2 contamination. For this, we will use the International Physical Activity Questionnaire (IPAQ).

SUMMARY:
The present study aims to assess the impact of exercise training, physical activity, and sedentary lifestyle on clinical outcomes in surviving patients infected with the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Therefore, this study will evaluate cross-sectionally and through a questionnaire in Portuguese and English on the internet, whether physically active patients have better outcomes for the disease such as shorter hospital stay, lesser symptoms, lesser need for mechanical ventilation, and medications.

DETAILED DESCRIPTION:
The new severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is responsible for the 2019 novel coronavirus (COVID-19) disease, initially discovered in the city of Wuhan, China, at the end of December 2019. In March 2020, the World Health Organization (WHO) declared SARS-CoV-2 as a worldwide pandemic. The disease quickly spread to several continents, also reaching Brazil strongly. This pandemic claimed (and still does) several victims, affecting more than 3 million confirmed cases worldwide with more than 200,000 deaths (official data: coronavirus.jhu.edu/map.html). In Brazil alone, by the time of writing this research project, 60,311 cases have been confirmed with 4,117 deaths. Epidemiological studies show that these numbers can be even higher, reaching up to eight times the number of cases.

As a new virus with such lethality and without the knowledge of its pathophysiology, WHO and the governments of each country have adopted isolation and social distance as a preventive measure to contain the spread of the virus, especially among the most vulnerable people such as the elderly, obese, diabetics and patients with cardiovascular diseases. So far, there is no effective and scientifically proven treatment for the disease, nor a vaccine for its effective control. In this sense, preventive measures such as personal hygiene, good nutrition and physical exercise seem to be the best forms of prevention. However, it is not known whether these measures can prevent contagion or whether they help the recovery of patients infected with SARS-CoV-2. It is well known that exercise training improves the response of the immune system providing protection against infections caused by intracellular microorganisms, thus being an important prevention strategy against SARS-CoV-2.

The present study aims to assess the impact of exercise training, physical activity, and sedentary lifestyle on clinical outcomes in surviving patients infected with the SARS-CoV-2 virus. Therefore, this study will evaluate cross-sectionally and through a questionnaire in Portuguese and English on the internet, whether physically active patients have better outcomes for the disease such as shorter hospital stay, lesser symptoms, lesser need for mechanical ventilation and medications.

ELIGIBILITY:
Inclusion Criteria:

* Men and women recovered and survivors of the disease
* With or without symptoms
* Patients with disease confirmation by reverse transcription-polymerase chain reaction (RT-PCR) test, blood test (serology), and a rapid antibody test
* With or without the need for hospitalization (nursery, semi-intensive and intensive unit)
* With or without the need for drug treatment
* Presence of any chronic disease such as diabetes, hypertension, coronary artery disease, obesity, metabolic syndrome, cancer, among others
* Literate patients in Portuguese and/or English.

Exclusion Criteria:

* Illiterate patients with difficulties in filling out the electronic form
* Patients still hospitalized and/or with symptoms of COVID-19

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surviving patients infected with SARS-CoV-2, as confirmed by a reverse transcription-polymerase chain reaction (RT-PCR) test, blood test (serology), and a rapid antibody test in Brazil and worldwide, will be considered eligible for the study. Only those patients fully recovered from the disease and asymptomatic will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1574 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Number of hospitalizations | Up to 6 months after hospital discharge and/or full recovery from the disease (asymptomatic)
  Number of hospitalizations required due to COVID-19

SECONDARY OUTCOMES:
Percentage of symptoms of the disease | Up to 6 months after hospital discharge and/or full recovery from the disease (asymptomatic)
  Symptoms such as fever, cough, shortness of breathe, and muscle pain due to COVID-19
Length of hospital stay | Up to 6 months after hospital discharge and/or full recovery from the disease (asymptomatic)
  Length of hospital stay required due to COVID-19
Percentage of mechanical ventilation | Up to 6 months after hospital discharge and/or full recovery from the disease (asymptomatic)
  Need for mechanical ventilation during hospitalization due to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo R Santos, PhD, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- Marcelo Rodrigues dos Santos, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared publicly through the tool Open Science Framework.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting in June 2020. All the data will be available permanently.
Access Criteria: Data will be available to other researchers after the end of the study. Data will be available for statistical analyses. The personal data of volunteers will not be identified. The principal investigator will be responsible for requests and criteria for information that will be shared.
URL: https://osf.io/crv6t/